CLINICAL TRIAL: NCT07384091
Title: The Diagnostic Accuracy of Ankle Audiometry Performed With the B250 for Superior Canal Dehiscence Syndrome in Patients Affected by Pulsatile Tinnitus and/or Autophony Disorders
Acronym: AA by B250
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Luca Verrecchia, Principal investigator, Region Stockholm
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2025-7292
Record Dates: First submitted 2026-01-20; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Superior Canal Dehiscence Syndrome; Autophony; Pulsatile Tinnitus
Keywords: SCDS; Ankle audiometry; B250
MeSH Terms: conditions — Semicircular Canal Dehiscence; Tinnitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ankle audiometry testing with B250 (Experimental): The arm consist of 30 consecutive adults (18-64 years) with autophony and/or pulsatile tinnitus, of which at least 15 are affected by superior canal dehiscense syndrome. All subjects will undergo testing with ankle audiometry (intervention) according to the method described in PMID: 36634643
  Interventions: Diagnostic Test: Ankle audiometry performed with the B250 transducer

INTERVENTIONS:
Diagnostic Test: Ankle audiometry performed with the B250 transducer — Calibrated vibration stimulation with a frequency of 250 Hz is applied at the ankle with the B250 transducer starting at an intensity of 80 dB FL. An incremental increase/decrease in the intensity of the applied bone vibration stimulus is employed in a manner similar to that performed during a standard pure tone hearing test. This is done in order to find the threshold in dB FL (at the ankle) for which the patient hears the sound in the target ear (right) is measured. The maximum applied intensity at the ankle will be 140 dB FL.

SUMMARY:
The goal of this clinical trial is to learn if the ankle audiometry test performed with the B250 bone conduction transducer can identify patients with superior canal dehiscence syndrome from those without among subjects presenting with autophony (a hearing condition where you hear your own body sounds) and/or pulsatile tinnitus.

The main question it aims to answer:

• Can ankle audiometry performed with B250 identify the condition of superior canal dehiscence syndrome among patients with autophony and/or pulsatile tinnitus, with a significance level of 80% and power level of 15%?

Study participants will undergo ankle audiometry testing with the B250 and the threshold in dB FL (at the ankle) for which the patient hears the sound in the target ear will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 64 years.
* Patients with symptoms of autophony and/or pulsatile tinnitus either due to a confirmed diagnosis of SCDS or not due to SCDS.

Exclusion Criteria:

* Severe sensorineural hearing.
* Middle ear or ear canal pathologies.
* Vulnerable patients.
* Confirmed intolerance or contraindication for body (ankle) vibratory stimulation.
* Anatomical body anomalies affecting normal testing procedure or interpretation of results.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The detection of SCDS among patients with autophony and/or pulsatile tinnitus. | At the end of the performed ankle audiometry test.

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska University Hospital, Hearing and Balance Unit, Stockholm, Huddinge, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ward BK, van de Berg R, van Rompaey V, Bisdorff A, Hullar TE, Welgampola MS, Carey JP. Superior semicircular canal dehiscence syndrome: Diagnostic criteria consensus document of the committee for the classification of vestibular disorders of the Barany Society. J Vestib Res. 2021;31(3):131-141. doi: 10.3233/VES-200004. PMID 33522990
- [Background] Verrecchia L, Freden Jansson KJ, Westin M, Velikoselskii A, Reinfeldt S, Hakansson B. Ankle Audiometry: A Clinical Test for the Enhanced Hearing Sensitivity for Body Sounds in Superior Canal Dehiscence Syndrome. Audiol Neurootol. 2023;28(3):219-229. doi: 10.1159/000528407. Epub 2023 Jan 12. PMID 36634643
- [Background] Watson SR, Halmagyi GM, Colebatch JG. Vestibular hypersensitivity to sound (Tullio phenomenon): structural and functional assessment. Neurology. 2000 Feb 8;54(3):722-8. doi: 10.1212/wnl.54.3.722. PMID 10680810